CLINICAL TRIAL: NCT03867240
Title: The Use of Perioperative Gabapentin in Adolescents Undergoing Posterior Spinal Fusion for Idiopathic Scoliosis to Prevent Chronic Postsurgical Pain, a Pilot Study.
Brief Title: Gabapentin and Chronic Post Surgical Pain
Acronym: CPSP
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study initially suspended recruitment due to COVID-19. Study withdrawn due to PI leaving institution in early 2021.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Cheryl Hartzell, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00106205
Record Dates: First submitted 2019-03-06; First posted 2019-03-07 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Pain, Postoperative; Scoliosis Idiopathic
Keywords: Gabapentin; Pain medication; Chronic postsurgical pain; Pediatric; Idiopathic scoliosis surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gabapentin (Experimental): Gabapentin is a common neuropathic medication used in the treatment of chronic pain. Gabapentin will be given preoperative and continued for 5 days postoperatively.
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): Control group will receive placebo medication at the same interval with the appropriate number of capsules or liquid for their weight to match the experimental group.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Gabapentin — Gabapentin (10 mg/kg up to 600 mg) will be given 30 minutes prior to being transported to the operating room. The gabapentin will be in the standard liquid with a concentration of 250mg/5mL. Starting postoperative day 1, patients in the experimental group will receive gabapentin three times daily. Dose of gabapentin will be 100 mg for patients <50 kg and 200 mg for patients > 50 kg. Gabapentin will be continued for 5 days postoperatively. If patients are discharged prior to postoperative day 5, they will be provided with gabapentin for the remainder of their doses upon discharge.
  Other Names: Neurontin
  Arms: Gabapentin
Other: Placebo — Placebo will be given 30 minutes prior to being transported to the operating room. Placebo will be identically appearing to gabapentin. Starting postoperative day 1, control group will receive placebo medication at the same interval with the appropriate number of capsules or liquid for their weight to match the experimental group. It will be continued for 5 days postoperatively. If patients are discharged prior to postoperative day 5, they will be provided with placebo for the remainder of their doses upon discharge.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the effect of a common pain medication (gabapentin) on chronic postsurgical pain in pediatric patients who require surgery for idiopathic scoliosis.

DETAILED DESCRIPTION:
Pain after surgery can last for a long time. When it lasts for over two months, it is considered chronic postsurgical pain (CPSP). This is a problem in kids and adolescents that can impact many areas of the patient's life and their family. Many patients who undergo surgery for their scoliosis develop CPSP. The purpose of this study is to investigate the effect of a common pain medication (gabapentin) on chronic postsurgical pain in pediatric patients who require surgery for idiopathic scoliosis.

ELIGIBILITY:
Inclusion Criteria:

* Be aged 10-18 years at the time of surgery
* Have a diagnosis of idiopathic scoliosis and/or kyphosis
* Be undergoing elective posterior spinal fusion
* Have only mild systemic disease

Exclusion Criteria:

* A diagnosis of neuromuscular scoliosis and/or kyphosis
* A diagnosis of chronic pain
* Used opioids in the past 6 months
* Developmental delay
* Liver or kidney disease
* Obstructive sleep apnea
* Body mass index >40
* Be pregnant or breastfeeding

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Change in NRS for pain intensity score comparing gabapentin and placebo groups | Baseline (prior to surgery), at 3 months postoperatively, and at 6 months postoperatively
  Patient's included in the study will rate their current pain using the numerical rating scale (NRS). With the NRS for pain intensity, the child rates their pain on a zero to 10 Likert scale, with zero being no pain and 10 being the most pain imaginable. A NRS > 4/10 at the time of the survey will be considered positive for CPSP.
Change in FDI score comparing gabapentin and placebo groups | Baseline (prior to surgery), at 3 months postoperatively, and at 6 months postoperatively
  The functional disability inventory (FDI) is a 15 question self-report inventory that assesses the impact of daily pain on activities at home, school, recreational and social domains. Items are rated on a five-point Likert Scale, ranging from 0 to 4, representing no trouble with the activity up to impossible to do the activity. The scores are tabulated, classifying the patient's function as no to minimal disability (0-12), moderate disability (12-29) or severe disability (30-60).

SECONDARY OUTCOMES:
Total narcotic requirement in the postoperative period in patients receiving gabapentin versus placebo | Postoperative period up to 1 month
  Opioid consumption will be tabulated from the postoperative care unit (PACU), across nursing shifts and cumulative amounts per day. IV morphine will be converted to oral morphine equivalents using a 3:1 ratio or IV hydromorphone will be converted to IV morphine using a 5:1 ratio. Oxycodone will be converted to oral morphine equivalents using a 1:1.5 ratio. All cumulative opioids will be reported as oral morphine equivalents.
Time to ambulation in patients receiving gabapentin versus placebo | Postoperative period up to 1 month
  Time to ambulation will be recorded.
First oral intake in patients receiving gabapentin versus placebo | Postoperative period up to 1 month
  Time to first oral intake will be recorded.
Time to discharge in each group in patients receiving gabapentin versus standard of care | Postoperative period up to 1 month
  Time to discharge will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Hartzell, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results after de-identification (text, tables, figures and appendices) will be shared. The following related documents will be available: study protocol, statistical analysis plan, analytic code. Data will become available immediately following publication and ending 5 years following article publication. Data will be shared with investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. Data will be shared for individual participant data meta-analysis. Request for proposal should be directed to Cheryl.maenpaa@emory.edu.To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will become available immediately following publication and ending 5 years following article publication.
Access Criteria: Data will be shared with investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose. Data will be shared for individual participant data meta-analysis.